CLINICAL TRIAL: NCT00057889
Title: A Phase II Open-Label Study of Single Agent MDX-010 for the Treatment of IL-2 Refractory or IL-2 Ineligible Patients With Stage IV Renal Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 030094; 03-C-0094; CDR0000285624; NCT00053729 (obsolete NCT alias)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Ipilimumab

INTERVENTIONS:
Biological: ipilimumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have metastatic renal cell cancer (kidney cancer) that is refractory to treatment with interleukin-2 or unable to be treated with interleukin-2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody in patients with metastatic clear cell renal cancer who are refractory to or ineligible for interleukin-2.
* Determine the impact of this drug on T-cell number and phenotype in these patients.

OUTLINE: This is an open-label study.

Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody IV over 90 minutes once every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with an ongoing partial response may receive additional courses of therapy.

Patients are followed at 4 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually until disease progression.

PROJECTED ACCRUAL: A total of 21-103 patients will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV clear cell renal carcinoma
* At least 1 site of measurable disease
* Meeting criteria for 1 of the following:

  * Disease progression after prior interleukin-2 (IL-2)
  * Ineligible for standard high-dose IV IL-2 due to comorbid medical conditions
  * Minimal disease (lesions ≤ 3 cm that do not pose risk to organ function) such that participation in this study is not likely to compromise the patient's opportunity to receive future high-dose IL-2
  * Indolent disease (defined as an increase in tumor size of < 50% within the past 6 months) such that participation in this study is not likely to compromise the patient's opportunity to receive future high-dose IL-2
  * No true papillary, medullary, chromophobe, collecting duct, or oncocytic renal cancer

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* WBC ≥ 2,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Hematocrit ≥ 30%

Hepatic

* AST ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ ULN (< 3.0 mg/dL for patients with Gilbert's syndrome)
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine < 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or any other cancer from which the patient has been disease free for at least 5 years
* No autoimmune disease (including uveitis and autoimmune inflammatory eye disease)
* No active uncontrolled infection
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody
* At least 3 weeks since prior immunotherapy for renal cancer

Chemotherapy

* At least 3 weeks since prior chemotherapy for renal cancer
* No concurrent chemotherapy

Endocrine therapy

* At least 3 weeks since prior hormonal therapy for renal cancer
* More than 4 weeks since prior corticosteroids
* No concurrent systemic or topical corticosteroids

Radiotherapy

* At least 3 weeks since prior radiotherapy for renal cancer

Surgery

* Not specified

Other

* Recovered from prior therapy
* At least 3 weeks since other prior therapy for renal cancer
* No concurrent immunosuppressive agents (e.g., cyclosporine and its analog)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Yang, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States